CLINICAL TRIAL: NCT06440902
Title: Exploration of Therapeutic Strategies for NeoRAS Wild-type Metastatic Colorectal Cancer Based on Circulating Tumor DNA: an Open, Prospective, Phase II Study
Brief Title: Exploration of Therapeutic Strategies for NeoRAS Wild-type Metastatic Colorectal Cancer Based on Circulating Tumor DNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ctDNA-neoRASCRC
Record Dates: First submitted 2024-02-22; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAS mutated metastatic colorectal cancer (Experimental): RAS mutated metastatic colorectal cancer were routinely treated after enrollment. When the disease progression was confirmed by imaging, peripheral blood ctDNA detection was performed to observe whether they were transformed into NeoRAS wild-type patients. If NeoRAS wild- type was detected, the anti-EGFR therapy may be considered as the following therapy for patients.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab is given In patients with NeoRAS WT
  Other Names: C225

SUMMARY:
Following systemic therapy in metastatic colorectal cancer(mCRC),RAS (including KRAS, NRAS and HRAS gene) status may change from a mutant(MT) to a wild-type(WT),a phenomenon known as "NeoRAS WT"mCRC.NeoRAS WT can be detected by longitudinal circulating tumor DNA(ctDNA) analysis.Therefore, this prospective phase II Study was design to explore the detection rate of peripheral blood ctDNA testing for NeoRAS WT and its guiding value for subsequent treatment for mCRC.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic colorectal cancer with tissue RAS mutation-type;
2. ECOG (Eastern Cooperative Oncology Group) performance score is 0-1;
3. Obtaining informed consent;
4. Surgical specimens or punctured tissue specimens containing tumors can be obtained; 10ml of peripheral blood can be obtained

Exclusion Criteria:

1. The pathology was not confirmed by colonoscopy biopsy or biopsy of metastasis;
2. Colorectal cancer patients with clinical stage I-III;Patients with RAS wild-type metastatic colorectal cancer confirmed by histological genetic testing;Lack of adequate organ functions, such as severe abnormalities in blood, liver and kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of NeoRAS WT | up to 60 months
  Proportion of occurrence of neoRAS WT

SECONDARY OUTCOMES:
Objective response rate(ORR) of NeoRAS wild-type patients receiving anti-EGFR therapy | Follow-up was conducted for 2 years after enrollment
  Objective response rate of NeoRAS wild-type patients receiving anti-EGFR (epidermal growth factor receptor) therapy
Progression-free survival (PFS) in NeoRAS WT patients | Follow-up was conducted for 2 years after enrollment
  Progression-free survival (PFS) : time from enrollment to disease progression from any cause
Overall survival (OS) in NeoRAS WT patients | Follow-up was conducted for 2 years after enrollment
  Overall survival (OS) : time from enrollment to death from any cause, loss of participants, and time of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Peng, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Osumi H, Takashima A, Ooki A, Yoshinari Y, Wakatsuki T, Hirano H, Nakayama I, Okita N, Sawada R, Ouchi K, Fukuda K, Fukuoka S, Ogura M, Takahari D, Chin K, Shoji H, Kato K, Ishizuka N, Boku N, Yamaguchi K, Shinozaki E. A multi-institutional observational study evaluating the incidence and the clinicopathological characteristics of NeoRAS wild-type metastatic colorectal cancer. Transl Oncol. 2023 Sep;35:101718. doi: 10.1016/j.tranon.2023.101718. Epub 2023 Jun 24. PMID 37364334
- [Background] Nicolazzo C, Magri V, Marino L, Belardinilli F, Di Nicolantonio F, De Renzi G, Caponnetto S, De Meo M, Giannini G, Santini D, Cortesi E, Gazzaniga P. Genomic landscape and survival analysis of ctDNA "neo-RAS wild-type" patients with originally RAS mutant metastatic colorectal cancer. Front Oncol. 2023 Mar 29;13:1160673. doi: 10.3389/fonc.2023.1160673. eCollection 2023. PMID 37064137
- [Background] Osumi H, Vecchione L, Keilholz U, Vollbrecht C, Alig AHS, von Einem JC, Stahler A, Striefler JK, Kurreck A, Kind A, Modest DP, Stintzing S, Jelas I. NeoRAS wild-type in metastatic colorectal cancer: Myth or truth?-Case series and review of the literature. Eur J Cancer. 2021 Aug;153:86-95. doi: 10.1016/j.ejca.2021.05.010. Epub 2021 Jun 18. PMID 34153718